CLINICAL TRIAL: NCT05075395
Title: Animal Assisted Interactions With an Animal Robot During Physical and Occupational Therapy Sessions in the Pediatric ICU: A Feasibility Study
Brief Title: Animal Assisted Interactions With Animal Robot in the Intensive Care Unit (ICU)
Acronym: PARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0005-19-EP
Record Dates: First submitted 2021-07-16; First posted 2021-10-12 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Critical Illness; Physical Therapy Modalities; Occupational Therapy; Animal Assisted Therapy
Keywords: Robot; Animal Assisted Interaction; Critical Care; Rehabilitation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): The Physical Therapy/Occupational Therapy (PT/OT) provider will assess whether the patient meets eligibility criteria. If the patient is eligible to participate, they will then introduce the study to the patient and their parent or guardian. If the patient is interested in participating, the PI or PI's research assistant (RA) will seek written informed consent. After informed consent is obtained, the PI or RA will begin pretest data collection. Then, the PT/OT provider will begin the therapy session with Paro. The PI or RA will remain in the room during therapy session to record field notes. When the therapy session is complete, the PI or RA will begin posttest data collection. The patient will remain in the study for up to 7 PT/OT sessions or until they are discharged from the PICU. The PT/OT providers will coordinate all subsequent therapy sessions with the PI/RA while the patient remains on the study protocol.
  Interventions: Device: PARO therapy seal

INTERVENTIONS:
Device: PARO therapy seal — PARO, a baby harp seal, is an advanced interactive, therapeutic medical robot developed by AIST, a leading Japanese industrial automation pioneer. It allows the documented benefits of animal therapy to be administered to patients in environments such as hospitals and extended care facilities where live animals present treatment or logistical difficulties.

SUMMARY:
The purpose of this study is to:

1. Establish the feasibility and acceptability of a therapeutic robot, Paro, for critically ill patients admitted to the Pediatric Intensive Care Unit
2. Explore safety considerations related to infection control [participant hospital-acquired infection (HAI) rates, screening for the presence of microbial contamination with real-time adenosine triphosphate (ATP) testing
3. Examine the therapeutic effect of Paro on patient psychological variables, physiological variables, and sedative and analgesic medication requirements.

DETAILED DESCRIPTION:
Admission to the Pediatric Intensive Care Unit (PICU) can be an extremely upsetting experience for children of all ages. In addition to physical symptoms such as pain, thirst and fatigue, patients in the PICU also experience a multitude of psychological symptoms. Symptoms like anxiety, spells of terror, social isolation, disturbed sleeping patterns, restlessness, fear, confusion and loss of control are exacerbated in the PICU because patients often have limited mobility, decreased capacity to communicate, and rely on healthcare providers for survival.

Large doses of sedative and analgesic medications are administered by nursing staff to help alleviate distressing symptoms. Overuse of sedative medications can cause a sequela of adverse effects, and therefore, recent recommendations call for reducing sedative use as much as possible. To minimize the overwhelming symptom burden of acute critical illness and promote lasting psychological well-being during recovery, it is imperative to identify effective non-pharmacological interventions that decrease psychological distress, but do not alter level of alertness during acute critical illness. Established evidence supports the use of a variety of non-pharmacological approaches that can be easily applied as adjuncts to sedative and analgesic medications in order to reduce dependence on these medications. Animal assisted interactions (AAI) are a promising integrative approach that can be used as an adjunct to sedative and analgesic medications in order to improve psychological symptoms and promote comfort, relaxation, and positive mood in critically ill patients.

AAI are interventions that intentionally incorporate animals as part of a therapeutic process to promote human health, learning, and well-being. Domestic and farm animals such as dogs, cats, birds, equines, guinea pigs, rabbits, llamas, sheep, goats, and pigs are predominantly featured in AAI programs. Animals can be simply observed, touched, held, and petted, or more actively integrated into specific therapy activities such as brushing with different tools to exercise range of motion and fine motor coordination and tandem walking with the animal to encourage exercise. Recent literature indicates that AAI can improve reality orientation and attention span, eliminate the sense of isolation, reduce stress and anxiety, enhance communication, promote positive social interactions, and enhance overall quality of life. The use of AAI in the ICU has the potential to engage patients, family members, and healthcare staff in an innovative, holistic approach to symptom management.

ELIGIBILITY:
Inclusion Criteria:

* age 5-18
* admitted to the PICU
* have an available parent or guardian
* an active consult request for physical therapy or occupational therapy
* awake, alert, and able to follow commands
* able to understand English
* free from significant vision or hearing deficits
* able to verbalize

Exclusion Criteria:

* have a pacemaker
* have droplet, enteric, or enhanced contact precautions
* have open wounds without a covering dressing or a dressing that is visibly soiled
* have known adverse psychological reactions to animals
* show signs of acute agitation (yelling, screaming, moaning, or is otherwise inconsolable)
* have excessive bodily secretions per primary bedside nurse
* report feeling nauseated

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Breanna Hetland, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: pediatric Intensive Care Unite (PICU) patients from a single tertiary medical center
Groups:
- Intervention: The Physical Therapy/Occupational Therapy (PT/OT) provider will assess whether the patient meets eligibility criteria. If the patient is eligible to participate, they will then introduce the study to the patient and their parent or guardian. If the patient is interested in participating, the PI or PIs research assistant (RA) will seek written informed consent. After informed consent is obtained, the PI or RA will begin pretest data collection. Then, the PT/OT provider will begin the therapy session with Paro. The PI or RA will remain in the room during therapy session to record field notes. When the therapy session is complete, the PI or RA will begin post-test data collection. The patient will remain in the study for up to 7 PT/OT sessions or until they are discharged from the Pediatric Intensive Care Unite (PICU). The PT/OT providers will coordinate all subsequent therapy sessions with the PI/RA while the patient remains on the study protocol.
  PARO therapy seal: PARO, a baby harp seal, is an advanced interactive, therapeutic medical robot developed by AIST, a leading Japanese industrial automation pioneer. It allows the documented benefits of animal therapy to be administered to patients in environments such as hospitals and extended care facilities where live animals present treatment or logistical difficulties.
Period: Overall Study
Arm/Group | Intervention
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: The PT/OT provider will assess whether the patient meets eligibility criteria. If the patient is eligible to participate, they will then introduce the study to the patient and their parent or guardian. If the patient is interested in participating, the PI or PIs research assistant (RA) will seek written informed consent. After informed consent is obtained, the PI or RA will begin pretest data collection. Then, the PT/OT provider will begin the therapy session with Paro. The PI or RA will remain in the room during therapy session to record field notes. When the therapy session is complete, the PI or RA will begin posttest data collection. The patient will remain in the study for up to 7 PT/OT sessions or until they are discharged from the PICU. The PT/OT providers will coordinate all subsequent therapy sessions with the PI/RA while the patient remains on the study protocol.
  PARO therapy seal: PARO, a baby harp seal, is an advanced interactive, therapeutic medical robot developed by AIST, a leading Japanese industrial automation pioneer. It allows the documented benefits of animal therapy to be administered to patients in environments such as hospitals and extended care facilities where live animals present treatment or logistical difficulties.
Arm/Group | Intervention
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.37 (3.905)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 4
  Caucasian | 11
  Hispanic | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Pain: Wrong-Baker FACES Pain Rating Scale [Mean (Standard Deviation); unit: Scores on a scale] — Population: Two participants did not complete the baseline measure for pain score
  Scores on a scale
    number analyzed (Participants) | 17
    (all) | 3.94 (3.455)
Children's Anxiety Meter-State (CAM-S) [Mean (Standard Deviation); unit: units on a scale] — State anxiety is anxiety at this moment in time. The measure is a vertical analog for child self-report of state. The CAM scale is drawn to resemble a thermometer with a bulb at the bottom and horizontal lines at intervals going up to the top. Children are instructed to Pretend that all of your worried or nervous feelings are in the bottom part of the thermometer. If you are a little bit worried or nervous, the feelings come up in the thermometer just a little bit. If you are very, very worried or nervous, the feelings go all the way to the top. The range is 0 to 10, 10 being the highest. Population: 3 participants did not complete the baseline score for anxiety
  units on a scale
    number analyzed (Participants) | 16
    (all) | 2.88 (2.419)
Physiologic Variables- Heart Rate [Mean (Full Range); unit: beats per minute] | 102 [69 to 129]
Physiologic Variables- Blood Pressure [Mean (Full Range); unit: Millimeters of mercury (mm Hg)]
  Systolic | 118 [98 to 151]
  Diastolic | 70 [55 to 83]
Physiologic Variables- Respiratory Rate [Mean (Full Range); unit: breaths per minute] | 22 [14 to 32]
Physiologic Variables- Oxygen [Mean (Full Range); unit: percentage of blood oxygen saturated] | 96 [91 to 99]

OUTCOME MEASURES:

1. Primary Outcome: Pain: Wrong-Baker FACES Pain Rating Scale
Description: The scale shows a series of faces ranging from a happy face at 0 which represents "no hurt" to a crying face at 10 which represents "hurts worst." Based on the faces and descriptions, the patient chooses the face that best describes their level of pain.
Time Frame: Baseline measures data recorded within ten minutes prior to the therapy session, outcome measure data recorded within ten minutes after each therapy session and an average of the after-therapy session scores was record.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 17
units on a scale | 3.94 (3.455)

2. Primary Outcome: Anxiety: Children's Anxiety Meter-State (CAM-S)
Description: The CAM scale is drawn to resemble a thermometer with a bulb at the bottom and horizontal lines at intervals going up to the top. Children are instructed to "Pretend that all of your worried or nervous feelings are in the very bottom down here. If you are a little bit worried or nervous, the feelings might come up just a little bit. If you are very, very worried or nervous, the feelings might go all the way to the top. Put a line showing how much worry or nervousness you feel." The range is 0 to 10 with 0 being no worry and 10 being the highest.
Time Frame: Baseline measures data recorded within ten minutes prior to the therapy session, outcome measure data recorded within ten minutes after each therapy session and an average of the after-therapy session scores was recorded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
units on a scale | 2.24 (2.700)

3. Primary Outcome: Hospital Acquired Infections- Central Lines
Description: Rates of Central Line Associated Blood Stream Infections (CLABSI) will be collected from the electronic medical record.
Time Frame: Chart review will be conducted staring the first day the participant is enrolled and continuing until 1 week after study completion. Participation varies for each participant between 1 and 7 sessions, depending on the length of ICU stay per participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants
  No Infection | 14
  Yes Infection | 1
  Unknown | 4

4. Primary Outcome: Hospital Acquired Infections- CAUTI
Description: Rates of Catheter-Associated Urinary Tract Infections (CAUTI) will be collected from the electronic medical record.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants
  No Infection | 15
  Unknown | 4

5. Primary Outcome: Hospital Acquired Infections- Enteroviruses
Description: Rates of Enteroviruses will be collected from the electronic medical record.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants
  No Infection | 15
  Unknown | 4

6. Primary Outcome: Hospital Acquired Infections- Influenza
Description: Rates Influenza will be collected from the electronic medical record.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants
  No Infection | 15
  Unknown | 4

7. Primary Outcome: Hospital Acquired Infections - Multi-drug-resistant Organisms (MDR) Organisms
Description: Rates of Multi-Drug Resistant Organisms will be collected from the electronic medical record.
Time Frame: as for outcome 3
Population: Intervention Group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants | 1

8. Primary Outcome: Hospital Acquired Infections- Surgical Site
Description: Surgical-Site Infections (SSI) will be collected from the electronic medical record.
Time Frame: as for outcome 3
Population: Intervention Group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants | 1

9. Primary Outcome: Hospital Acquired Infections- VAP
Description: Rates of Ventilator-Associated Pneumonia (VAP) will be collected from the electronic medical record.
Time Frame: as for outcome 3
Population: Intervention Group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants | 1

10. Primary Outcome: Microbial Contamination Screening
Description: The Adenosine triphosphate (ATP) Monitoring with SystemSURE Plus Process uses a process which monitors levels of ATP Bioluminescence. We will implement an established cleaning protocol and then measure ATP after a PT/OT session by swabbing PARO on the following areas: head, right flipper, left flipper, bottom [by on/off switch], top left back area, top right back area, stomach [underneath]. Relative Light Units were averaged across all regions to get one measure per participant. The amount of bioluminescence is measured by the luminometer and the result is given in units known as the relative light units. The ATP bioluminescence reaction is linear, the more ATP present means the more light will be present. The measure of ATP can therefore be determined indirectly by determining the measure of Rlu in living organisms and even organic materials.
Time Frame: Screen was completed immediately after each individual session on the PARO and an average was reported
Population: Intervention Group
Measure: Mean (Standard Deviation); unit: Relative Light Units (RLU)
Arm/Group | Intervention
Number analyzed (Participants) | 19
Relative Light Units (RLU) | 7 (4.8)

11. Primary Outcome: Activity Performance Form
Description: The Activity Performance Form is an investigator developed measure that assesses the length of each therapy session (in minutes).
Time Frame: Outcome measure data recorded within ten minutes after the therapy session has ended
Measure: Mean (Standard Deviation); unit: Minutes per session
Arm/Group | Intervention
Number analyzed (Participants) | 19
Minutes per session | 35.8 (9.7)

12. Primary Outcome: Physiologic Variables- Heart Rate
Description: Measure heart Rate before and after therapy session
Time Frame: Baseline measures data recorded within ten minutes prior to the therapy session, outcome measure data recorded within ten minutes after each therapy session and an average of the after-therapy session score was recorded.
Measure: Mean (Full Range); unit: beats per minute
Arm/Group | Intervention
Number analyzed (Participants) | 19
beats per minute | 99 [55 to 128]

13. Primary Outcome: Physiologic Variables- Blood Pressure
Description: Measure blood pressure before and after each session.
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: millimeters of mercury (mmHg)
Arm/Group | Intervention
Number analyzed (Participants) | 19
millimeters of mercury (mmHg)
  Systolic BP - Post | 119 [104 to 139]
  Diastolic BP- Post | 71 [59 to 89]

14. Primary Outcome: Physiologic Variables- Respiratory Rate
Description: Measure respiratory rate before and after each session.
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: breaths per minute
Arm/Group | Intervention
Number analyzed (Participants) | 19
breaths per minute | 25 [14 to 40]

15. Primary Outcome: Physiologic Variables- Oxygen
Description: Measure oxygen saturation before and after each session.
Time Frame: Baseline measures show data recorded within ten minutes prior to the therapy session, outcome measure shows data recorded within ten minutes after the therapy session and an average of the after therapy session scores was recorded.
Measure: Mean (Full Range); unit: percent of blood cells saturated
Arm/Group | Intervention
Number analyzed (Participants) | 19
percent of blood cells saturated | 97 [92 to 100]

ADVERSE EVENTS:
Time Frame: Adverse event data was recorded for up to 7 sessions or discharge from the Pediatric ICU, whichever comes first; for an average of 2.5 sessions.
Description: We did not use a different definition of adverse event from the ClinicalTrials.gov definitions.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT05075395/Prot_SAP_006.pdf
  • Informed Consent Form (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT05075395/ICF_005.pdf